CLINICAL TRIAL: NCT07342881
Title: A Phase 1 Non-Randomized, Open-Label, Single Dose Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Pevifoscorvir Sodium (ALG-000184) in Participants With Renal Impairment and in Healthy Participants With Normal Renal Function
Brief Title: Single Dose Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Pevifoscorvir Sodium (ALG-000184) in Participants With Renal Impairment and in Healthy Participants With Normal Renal Function
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aligos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALG-000184-208
Record Dates: First submitted 2025-12-15; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Chronic Hepatitis B Infection
Keywords: Chronic Hepatitis B Infection
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Intervention Model Description: This is a Phase 1 non-randomized, open-label, single-dose study of pevifoscorvir sodium (also known as ALG-000184) in participants with severe renal impairment (Part 1), in participants with mild or moderate renal impairment (Optional Part 2) and in participants without renal impairment (Parts 1 and 2), matched for age, body weight and, to the extent possible, for sex.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Subjects with renal Impairment (Experimental): Subjects with renal impairment will receive single oral doses of 100 mg pevifoscorvir sodium. Subjects will be followed up for 14 days after the administration of study drug.
  Interventions: Drug: Pevifoscorvir Sodium (ALG-000184)
- Subjects without renal impairment (Experimental): Subjects without renal impairment will receive single oral doses of 100 mg pevifoscorvir sodium. Subjects will be followed up for 14 days after the administration of study drug.
  Interventions: Drug: Pevifoscorvir Sodium (ALG-000184)

INTERVENTIONS:
Drug: Pevifoscorvir Sodium (ALG-000184) — Pevifoscorvir Sodium (ALG-000184) Single oral doses of 100 mg pevifoscorvir sodium

SUMMARY:
This is a Phase 1 non-randomized, open-label, single-dose study of pevifoscorvir sodium (also known as ALG-000184) in participants with severe renal impairment (Part 1), in participants with mild or moderate renal impairment (Optional Part 2) and in participants without renal impairment (Parts 1 and 2), matched for age, body weight and, to the extent possible, for sex.

ELIGIBILITY:
Inclusion Criteria for All Subjects:

1. Male and Female between 18 and 75 years old
2. Body Mass Index (BMI) 17.5 to 40.0 kg/m^2 and a total body weight >50 kg (110 lb)
3. Female subjects must either be not of childbearing potential or if they are a woman of childbearing potential, they are only eligible if they and any non-sterile, male sexual partners agree to use highly effective contraceptive therapy

Inclusion Criteria for Subjects with Normal Renal Function:

1. Good general health as defined by no clinically relevant abnormalities identified by Medical History and a vital signs, clinical laboratory and 12-lead electrocardiogram (ECG) assessment
2. Subjects must fit the demographic-matching criteria including body weight, age, and to the extent possible, sex
3. Normal renal function (estimated Glomerular Filtration Rate [eGFR] ≥90 mL/min) with no known or suspected renal impairment

Inclusion Criteria for Subjects with Impaired Renal Function:

1. Subject satisfies the eGFR criteria for renal impairment classification within 28 days of study drug administration
2. Any form of renal impairment except acute nephritic syndrome (subjects with history of previous nephritic syndrome but in remission can be included).
3. Stable concomitant medications for the management of an individual subject's medical history for at least 28 days prior to screening
4. Subjects must have a 12-lead ECG and vital signs assessment that meet the protocol criteria

Exclusion Criteria for All Subjects:

1. Subjects with any current or previous illness that, in the opinion of the Investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject or that could prevent, limit, or confound the protocol specified assessments or study results and interpretation
2. Subjects with a past history of cardiac arrhythmias, risk factors for Torsade de Pointes syndrome (e.g., hypokalemia, family history of long QT Syndrome) or recent history or clinical evidence at screening of significant (subjects with normal renal function) or unstable (subjects with renal impairment) cardiac disease etc.
3. Subjects with a history of clinically significant drug allergy
4. Subjects with a recent (within 1 year of randomization) history or current evidence of drug abuse or recreational drug use
5. Excessive use of alcohol defined as regular consumption of ≥14 units/ week for women and ≥21 units/week for men
6. Unwilling to abstain from alcohol use for 48 hours prior to start of the study through end of study follow up
7. Subjects with Hepatitis A, B, C, E or HIV-1/HIV-2 infection or acute infections such as SARS- CoV-2 infection
8. Subjects with alanine aminotransferase (ALT) or aspartate aminotransferase (AST) values >2x upper limit of normal (ULN)
9. Subjects with bilirubin (total, direct) >1.5x ULN (unless Gilbert's is suspected)
10. Positive pregnancy test; females must not be pregnant at enrollment

Exclusion Criteria for Subjects with Normal Renal Function:

1. Hemoglobin <10 g/dL

Exclusion Criteria for Subjects with Impaired Renal Function:

1. Participants requiring hemodialysis and/or peritoneal dialysis
2. Hemoglobin <9 g/dL

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration time curve [AUC] | Up to 4 days
  Plasma PK parameters in each cohort of total ALG-001075 and the metabolite ALG-000302
Maximum plasma concentration [Cmax] | Up to 4 Days
  Plasma PK parameters in each cohort of total ALG-001075 and the metabolite ALG-000302
Minimum plasma concentration [Cmin] | Up to 4 Days
  Plasma PK parameters in each cohort of total ALG-001075 and the metabolite ALG-000302
C0 [predose] | Up to 4 days
  Plasma PK parameters in each cohort of total ALG-001075 and the metabolite ALG-000302
Half-life [t1/2] | Up to 4 Days
  Plasma PK parameters in each cohort of total ALG-001075 and the metabolite ALG-000302
Time to maximum plasma concentration [Tmax] | Up to 4 Days
  Plasma PK parameters in each cohort of total ALG-001075 and the metabolite ALG-000302
Apparent Clearance (CL/F) | Up to 4 Days
  Plasma PK parameters in each cohort of total ALG-001075 and the metabolite ALG-000302
Apparent Volume of Distribution (V/F) | Up to 4 Days
  Plasma PK parameters in each cohort of total ALG-001075 and the metabolite ALG-000302
Total Amount of Drug Excreted in Urine (Ae) | Up to 4 Days
  Urine PK parameters in each cohort of total ALG-001075 and the metabolite ALG-000302
Renal Clearance (CLr) | Up to 4 Days
  Urine PK parameters in each cohort of total ALG-001075 and the metabolite ALG-000302

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 15 days
  The number and severity of treatment emergent events in subjects with renal impairment and subjects with normal renal function as assessed by DAIDS v2.1

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Orlando Clinical Research Center, Orlando, Florida
  - Genesis Clinical Trials, Tampa, Florida